CLINICAL TRIAL: NCT00832559
Title: A Phase I, Open-label, Dosage Escalation, Study of Multiple Doses of CAVATAKTM (CVA21; Coxsackievirus A21) Administered Intratumourally in the Treatment of Squamous Cell Carcinoma of the Head and Neck Bearing ICAM-1 Receptors (VLA-X06)
Brief Title: A Study of the Intratumoural Administration of CAVATAK to Head and Neck Cancer Patients (VLA-X06)
Acronym: VLA-X06
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor recruitment rate.
Sponsor: Viralytics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V937-005; VLA-X06/PSX-X06 (Other: Viralytics Study ID)
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Head and Neck Cancer
Keywords: CAVATAK; Coxsackievirus A21; CVA21; Oncolytic virotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

ARMS (1):
- CVA21 (Experimental): CVA21
  Interventions: Biological: CVA21

INTERVENTIONS:
Biological: CVA21 — 1, 3 or 6 doses of CAVATAK (10^9 TCID50) at 48 hour intervals.
  Other Names: CAVATAK; Coxsackievirus A21

SUMMARY:
This study is designed to assess the safety and initial indications of efficacy resulting from multiple doses of CAVATAK injected directly into solid tumours of the Head and Neck that have been confirmed to express ICAM-1 and DAF.

CAVATAK (Coxsackievirus A21) is a naturally occurring common cold virus that preclinical research indicates can preferentially infect and kill cancer cells expressing the receptors ICAM-1 and/or DAF. This virus is known to cause self limiting upper respiratory infections and has been used previously to challenge therapies against the common cold. The virus is not generically modified.

The study proposes to administer CAVATAK to three cohorts each of three patients. The first cohort will receive a single dose, the second cohort will receive three doses, and the final cohort will receive six doses. There will a 48 hour interval between repeated doses.

The primary objective of the study is to determine the safety and efficacy of CVA21 given by intratumoural injection in the treatment of recurrent, unresectable squamous cell carcinoma of the head and neck by measuring primary and field tumour status and adverse effects.

Secondary objectives of the study are:

1. Indirect measurements of efficacy by measuring appropriate biomarkers in serum and tumour biopsy samples for viral replication, induction of apoptosis and anti-tumour immune responses.
2. To determine the time course of potential primary and secondary viraemia.
3. To characterise the time course of the anti-CVA21 antibody response after administration of CVA21

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are willing and able to provide written informed consent to participate in the study.
2. Patients with histologically confirmed metastatic or recurrent squamous cell carcinoma of the head or neck currently documented as "progressive disease"
3. Head and neck cancer patients with at least one tumour mass where the tumour mass is accessible for intratumoural injection and can be measured at periodic intervals for tumour size using callipers and/or ultrasound.
4. All patients to have histologically confirmed squamous cell carcinoma of the head and neck (excluding nasopharyngeal) that had recurred or relapsed after surgery and/or radiotherapy and/or chemotherapy.
5. The longest diameter of the target injectable tumour being no greater than 6 cm or no less than 1 cm in the longest diameter.
6. The tumour mass to be intratumourally injected to be easily accessible for injection and amenable to measurement by physical examination and / or radiographically.
7. Patients to be 18 years or older
8. Absence of circulating antibodies to CVA21 (titre < 1:16).
9. Adequate haematological, hepatic and renal function, defined as:

   ANC > 1.5 x 109/L, platelets > 100 x 109/L Bilirubin < 20µmol/L, AST < 2.5 times the upper limit of normal Calculated creatinine clearance > 30 mL/minute

   Adequate immunologic function, defined as:

   Serum IgG > 5g/L T cell subsets within normal limits
10. Fertile males and females must agree to the use of an adequate form of contraception. Hormonal contraceptives should be supplemented with an additional barrier method. Negative pregnancy test is required in female patients of child-bearing potential.

Exclusion Criteria:

1. Patients receiving radiotherapy to the proposed injected tumour or radiotherapy within the last 3 weeks
2. Performance status > 1 on the ECOG scale
3. Life expectancy < 3 months.
4. Pregnancy or breastfeeding.
5. Primary or secondary immunodeficiency, including immunosuppressive disease, and immunosuppressive doses of corticosteroids (e.g. prednisolone > 7.5mg per day) or other immunosuppressive medications including cyclosporine, azathioprine, interferons, within the past 4 weeks.
6. Positive serology for HIV, Hepatitis B or Hepatitis C.
7. Splenectomy.
8. Presence of uncontrolled infection.
9. Any uncontrolled medical condition that in the opinion of the Investigator is likely to place the patient at unacceptable risk during the study or reduce their ability to complete the study
10. Participation in another study requiring administration of an investigational drug or biological agent within the last 4 weeks
11. Known allergy to treatment medication or its excipients
12. Tumours to be injected lying in mucosal regions or close to an airway, major blood vessel or spinal cord that, in the opinion of the Investigators, could cause occlusion or compression in the case of tumour swelling or erosion into a major vessel in the case of necrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-01-27 (Actual); Primary Completion 2011-07-28 (Actual); Study Completion 2011-07-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of patients to multiple doses of CAVATAK | 1 year
  safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ackland, MBBS FRACP, Principal Investigator — Principal Investigator
Locations (3):
- Australia (3):
  - St Vincents Hospital, Darlinghurst, New South Wales
  - Calvary Mater Newcastle Hospital, Newcastle, New South Wales
  - Monash Medical Centre, Clayton, Victoria